CLINICAL TRIAL: NCT03445572
Title: Feasibility Study of Meditative Practices in Hospitalized Cancer Patients
Brief Title: Meditative Slow Breathing or Isha Kriya Meditation in Improving Cancer-Related Symptoms in Hospitalized Participants With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2017-0694; NCI-2018-00927 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2017-0694 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2018-02-19; First posted 2018-02-26 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-08

CONDITIONS: Malignant Neoplasm
MeSH Terms: conditions — Neoplasms | interventions — Practice Guidelines as Topic; Standard of Care; Meditation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I (MSB) (Experimental): Participants are instructed on the MSB technique and then perform MSB over 15 minutes BID for 28 days.
  Interventions: Procedure: Meditation Therapy; Other: Questionnaire Administration
- Group II (IK meditation) (Experimental): Participants are instructed on the 3 steps of IK meditation and then perform IK meditation over 15 minutes BID for 28 days.
  Interventions: Procedure: Meditation Therapy; Other: Questionnaire Administration
- Group III (waitlist) (Active Comparator): Participants are placed on a waitlist and receive standard supportive care for 28 days. After 28 days, participants may crossover to Group II.
  Interventions: Other: Best Practice; Other: Questionnaire Administration

INTERVENTIONS:
Other: Best Practice — Receive standard supportive care
  Other Names: standard of care; standard therapy
  Arms: Group III (waitlist)
Procedure: Meditation Therapy — Perform MSB
  Other Names: Meditation
  Arms: Group I (MSB)
Procedure: Meditation Therapy — Perform IK meditation
  Other Names: Meditation
  Arms: Group II (IK meditation)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This trial studies how well meditative slow breathing or Isha Kriya meditation works in improving cancer-related symptoms in hospitalized participants with cancer. Meditative slow breathing or Isha Kriya meditation may help to decrease perceived stress and enhance well-being in hospitalized cancer participants.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Test the feasibility of the meditation practice.

SECONDARY OBJECTIVES:

I. Explore the acceptability of meditation in cancer patients through modified Global Symptom Evaluation (GSE) and on day 7 +/- 1 day and day 28 +/- 3 days.

II. Explore the effect of meditative practices in cancer patients through Edmonton Symptom Assessment Scale (ESAS) on the day of enrolment and a weekly basis until the end of study at four weeks.

OUTLINE: Participants are randomized to 1 of 3 groups.

GROUP I (MSB): Participants are instructed on the meditative slow breathing (MSB) technique and then perform MSB over 15 minutes twice daily (BID) for 28 days.

GROUP II (IK MEDITATION): Participants are instructed on the 3 steps of Isha Kriya (IK) meditation and then perform IK meditation over 15 minutes BID for 28 days.

GROUP III (WAITLIST): Participants are placed on a waitlist and receive standard supportive care for 28 days. After 28 days, participants may crossover to Group II.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of malignancy
* Admitted to the hospital
* Able to follow instructions
* Eastern Cooperative Oncology Practice (Eastern Cooperative Oncology Group [ECOG]) score of 3 or below
* Fluency in English

Exclusion Criteria:

* Patients with life expectancy less than 2 months per attending physician or advance practice provider's note or assessment of prognosis
* Patients with cognitive dysfunction
* Patients who are admitted for observation for < 48 hours will be excluded from the study, as one day would be difficult to provide the necessary information
* Patients who are delirious
* Patients who are unable to follow instructions due to their medical condition
* Patients admitted to the intensive care unit
* Patients with ESAS > 4/10 on dyspnea
* Patients requiring oxygen more than 2 liters
* Patients who are current meditation practitioners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2018-09-21 (Actual); Primary Completion 2020-08-04 (Actual); Study Completion 2020-08-04 (Actual)

PRIMARY OUTCOMES:
Feasibility of the Meditation Practice defined by Recruitment Rate | Day 7
Feasibility of the Meditation Practice defined by Adherence Rate | Day 7

SECONDARY OUTCOMES:
Acceptability of Meditation in Cancer Patients Assessed by Modified Global Symptom Evaluation (GSE) | Day 7 and Day 28
Effect of Meditative Practices in Cancer Patients Assessed by Edmonton Symptom Assessment Scale (ESAS) | Enrollment and a weekly basis until the end of study at four weeks.
  Scale is from 0 to 10 with 0 being no symptoms to 10 being worse symptoms.
  Proportions of participants who consider that the study makes their symptoms better estimated along with a 90% confidence interval for each of the intervention groups. The Linear mixed model used to examine the differential changes over time for ESAS scores among the three groups.

CONTACTS AND LOCATIONS:
Overall Officials: Santhosshi Narayanan, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Narayanan S, Reddy A, Lopez G, Liu W, Wu J, Liu D, Manzano J, Williams JL, Mallaiah S, George M, Amaram J, Subramaniam B, Cohen L, Bruera E. Randomized Feasibility Study of Meditative Practices in Hospitalized Cancer Patients. Integr Cancer Ther. 2020 Jan-Dec;19:1534735420909903. doi: 10.1177/1534735420909903. PMID 32153208
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org